CLINICAL TRIAL: NCT02298803
Title: QT Interval Abnormalities in Sulfonylurea Treated Type 2 Diabetes: Relationship to Treatment Induced Hypoglycaemia and Glycaemic Variability Determined by Simultaneous Ambulatory Monitoring
Brief Title: QT Interval Abnormalities in Sulfonylurea Treated Type 2 Diabetes: Relationship to Treatment Induced Hypoglycaemia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Royal Prince Alfred Hospital, Sydney, Australia (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Dr Ted Wu, Principal Investigator, Royal Prince Alfred Hospital, Sydney, Australia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: X14 0314
Record Dates: First submitted 2014-11-18; First posted 2014-11-24 (Estimated); Results first posted 2018-02-28 (Actual); Last update posted 2018-02-28 (Actual); Status verified 2018-01

CONDITIONS: Diabetes Related Complications
MeSH Terms: conditions — Diabetes Complications

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Holter and Glucose monitoring (Other): In this study the interventions will be the simultaneous monitoring of glucose and QT interval via a subcutaneous continuous glucose monitor and a Hoter monitor, respectively.
  Interventions: Device: Holter and Glucose monitoring

INTERVENTIONS:
Device: Holter and Glucose monitoring — (i) Continuous Glucose Monitoring A sterile disposable glucose-sensing sensor will be inserted into the subcutaneous tissues in either the abdomen or the upper outer quadrant of the patient's buttock. This sensor automatically measures the change in glucose in interstitial fluid every 5 minutes. The monitor will be worn for two days.
  (ii)Holter Monitoring The Holter monitor to capture cardiac conduction, specifically QT interval, will be worn for the same period as the continuous glucoe monitor with study participants encouraged to perform regular daily activities.

SUMMARY:
Hypoglycaemia is the most common acute complication of diabetes and can limit therapeutic efforts to improve glycaemic control. It is a potential side effect of drugs used to treat diabetes, particularly with the use of sulfonylurea (SU) treatment. It has been demonstrated that hypoglycaemia causes the prolongation of corrected QT (QTc) interval, which is associated with ventricular arrhythmias and sudden death. Hypoglycaemia in T2DM has recently come into focus with the results of the ACCORD, ADVANCE and VADT trials.

In this study, the investigators aim to examine the association of hypoglycaemia and glucose fluctuations on QT-interval and QT variability in patients with type 2 diabetes treated with SU. Patients will be studied using simultaneous Continuous Glucose Monitoring (CGM) and ambulatory ECG monitoring (Holter).

Study participants will be recruited from the Diabetes Centre, RPAH or from specialist consulting rooms. They will be required to attend the Diabetes Centre on two occasions.

At the first visit, blood will be collected and CGM and Holter monitoring commenced. At Visit 2, i.e. two days later, the patient will return to the Diabetes Centre to have the equipment removed. The data obtained from the CGM and Holter monitor will then be downloaded for review and analysis.

DETAILED DESCRIPTION:
Background/Scientific Basis:

Hypoglycaemia is the most common acute complication of diabetes and can limit therapeutic efforts to improve glycaemic control. It is a potential side effect of the drugs used to treat diabetes, particularly with the use of exogenous insulin or insulin secretagogues, such as sulfonylurea (SU) treatment. As many people are prescribed these agents, hypoglycaemia is frequent in clinical practice, particularly as treatment targets have become more stringent. Several studies have demonstrated that insulin-induced hypoglycaemia causes prolongation of corrected QT (QTc) interal (Chugh et al), which is associated with ventricular arrhythmias and sudden death, perhaps as a result of hypokalaemia and an increase in serum catecholamines. Cardiac effects of hypoglycaemia are usually associated with type 1 diabetes and insulin therapy. Hypoglycaemia in type 2 diabetes (T2DM) on oral agents has not, until recently, been considered to be as serious. Recently, hypoglycaemia in T2Dm has come in into focus since the salutary results of the ACCORD, ADVANCE and VADT trails, each of which implicated hypoglycaemia as a cause for increased death. The majority of excess deaths in the intensive treatment group of ACCORD were classified as sudden cardiac death. There is now a growing body of evidence that hypoglycaemia is a pro-arrhythmic event via QT prolongation and particularly in the context of myocardial ischemia which reduces the tolerance of myocardial tissue for the further pro-arrhythmic action of hypoglycaemia.

It is notable that hypoglycaemia occurs commonly in those using SU. For example in the UK Hypoglycaemia Study (UK Hypoglycaemia Study Group) , 7% of individuals treated with SUs had at least one episode of severe (requiring external assistance) hypoglycaemia and the proportion reporting at least one mild (symptomatic, self-treated) episode was 39%, a rate comparable to insulin treatment. Furthermore, the SU receptor functions as the regulatory subunit of the adenosine triphosphate (ATP)-sensitive potassium (KATP) channel. KATP channels are widely expressed in the heart and vascular smooth muscle cells. There have been long-held concerns that SU effects on these channels may affect ischaemic preconditioning (Cleveland et al), a protective mechanism in the myocardium. This may represent an additive deleterious impact specific to SUs in a hypoglycaemic setting.

Despite these theoretical concerns associated with SU treatment the pro-arrhythmic effects of SU induced hypoglycaemia have not previously been easy to study in ambulatory patients. Now the dual ambulatory technologies of CGMS (Maia et al) and ambulatory ECG (Holter) monitoring provide an opportunity to examine this potential association under real life conditions. Even in the absence of absolute QT prolongation, there is evidence that beat-to-beat QT variability is also a risk marker for sudden death and ventricular arrhythmia (Piccirillo et al). Additionally, glucose variability may also have an impact on cardiac tissue. Habituation to chronic hyperglycaemia could lead to a situation where a sudden decrease to plasma glucose leads to changes in QT interval, even when the glucose falls within the normal range ("relative hypoglycaemia").

A pilot study in our institution of 14 individuals on insulin (3 with T1DM and 11 with T2DM) showed statistically significant prolongation of QTc during periods of hypoglycaemia. The mean difference in QTc during hypos was 7.8ms (p<0.05). An inverse relationship between the magnitude of increase in QTs during hypoglycaemia and baseline QTc was found. The limitations of the pilot study are that it was restricted to those subjects treated with insulin and that relative hypoglycaemia and QT variability were not analysed.

Hypothesis:

Sulfonylurea induced hypoglycaemia and/or fluctuations in glucose are pro-arrhythmic by prolonging the QTc interval and/or increasing beat-to-beat QTc variability. It is expected that the QT interval will be significantly longer during the hypoglycemic periods compared to the non-hypoglycemic periods in patients in T2DM treated with SU.

Aims:

To examine the association of hypoglycaemia and glucose fluctuations on QT-interval and QT variability in patients with type 2 diabetes treated with SU. Patients will be studied using simultaneous Continuous Glucose Monitoring (CGM) and ambulatory ECG monitoring (Holter).

Potential Significance:

The information gained from this study has the potential to improve our understanding of the relationship between hypoglycaemia and cardiac arrhythmia in patients with diabetes.

Recruitment Process:

Patients with type 2 diabetes attending the Diabetes Centre, Royal Prince Alfred Hospital who fulfils the entry criteria will be approached to participate in this study. They will be approached either when they attend the Diabetes Centre for treatment, or by means of a telephone call. The requirements of the study will be discussed with each potential participant and they will be given a copy of the Participant Information Sheet and Consent Form to take home and read. The proposed number of participants for this study is approximately 30 individuals.

Research Interventions:

1. Blood Collection
2. Continuous Glucose Monitoring
3. Home Blood Glucose Monitoring
4. Holter Monitor

Risk and Side Effects:

We do not anticipate any adverse events associated with study participation. However, there may be some mild discomfort and/or bruising at the site of blood collection, or insertion of the glucose sensor for CGM, or skin irritation from the ECG adhesive tapes required for Holter monitoring.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes
* A history of symptomatic or documented hypoglycaemia
* Currently treated with a sulphonylurea ± any anti-diabetic agent/s other than insulin
* Currently performing home blood glucose monitoring and willing to do seven tests a day during the study period

Exclusion Criteria:

* Type 1 diabetes
* Current treatment with insulin
* LBBB and conduction anomalies that preclude QT analysis
* Drugs that prolong QT interval
* Family history of Long QT syndrome

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2015-01; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ted Wu, MBBS, PhD, Principal Investigator — Royal Prince Alfred Hospital, Sydney, NSW, Australia

REFERENCES:
- [Background] Chugh SS, Reinier K, Singh T, Uy-Evanado A, Socoteanu C, Peters D, Mariani R, Gunson K, Jui J. Determinants of prolonged QT interval and their contribution to sudden death risk in coronary artery disease: the Oregon Sudden Unexpected Death Study. Circulation. 2009 Feb 10;119(5):663-70. doi: 10.1161/CIRCULATIONAHA.108.797035. Epub 2009 Jan 26. PMID 19171855
- [Background] UK Hypoglycaemia Study Group. Risk of hypoglycaemia in types 1 and 2 diabetes: effects of treatment modalities and their duration. Diabetologia. 2007 Jun;50(6):1140-7. doi: 10.1007/s00125-007-0599-y. Epub 2007 Apr 6. PMID 17415551
- [Background] Cleveland JC Jr, Meldrum DR, Cain BS, Banerjee A, Harken AH. Oral sulfonylurea hypoglycemic agents prevent ischemic preconditioning in human myocardium. Two paradoxes revisited. Circulation. 1997 Jul 1;96(1):29-32. doi: 10.1161/01.cir.96.1.29. PMID 9236412
- [Background] Maia FF, Araujo LR. Efficacy of continuous glucose monitoring system (CGMS) to detect postprandial hyperglycemia and unrecognized hypoglycemia in type 1 diabetic patients. Diabetes Res Clin Pract. 2007 Jan;75(1):30-4. doi: 10.1016/j.diabres.2006.05.009. Epub 2006 Jun 27. PMID 16806560
- [Background] Piccirillo G, Rossi P, Magri D. The QT variability index: a multidimensional approach to understanding cardiovascular disease. Cardiology. 2011;118(1):42-4. doi: 10.1159/000324476. Epub 2011 Mar 11. No abstract available. PMID 21411996

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients with type 2 diabetes attending the Diabetes Centre, Royal Prince Alfred Hospital who fulfilled the entry criteria were approached to participate. The requirements of the study were discussed and participants were given a copy of the Participant Information Sheet and Consent Form to read. 30 individuals were recruited in 2015.
Pre-assignment Details: 30 participants were screened and enrolled. Data from all 30 participants was included in the analysis.
Groups:
- Holter and Glucose Monitoring: In this study all participants underwent simultaneous monitoring of glucose and QT interval via a subcutaneous continuous glucose monitor and a Hoter monitor, respectively.
  Holter and Glucose monitoring: (i) Continuous Glucose Monitoring A sterile disposable glucose-sensing sensor was inserted into the subcutaneous tissue in the abdomen of the patient. This sensor automatically measured the average glucose concentration in interstitial fluid every 5 minutes. The monitor was worn for 48 hours.
  (ii)Holter Monitoring The Holter monitor was worn for the same period as the continuous glucose monitor. QT intervals were extracted using proprietary software. Study participants were encouraged to perform regular daily activities during monitoring.
Period: Overall Study
Arm/Group | Holter and Glucose Monitoring
Started | 30
Completed | 30
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Hypoglycemic Group: N=9; these participants experienced at least one episode of hypoglycaemia (blood glucose level <3.5mmol/L) during the monitoring period.
- Normoglycemic Group: N=21; these participants experienced no episodes of hypoglycaemia during the monitoring period.
- Total: Total of all reporting groups
Arm/Group | Hypoglycemic Group | Normoglycemic Group | Total
Number analyzed (Participants) | 9 | 21 | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.8 (10.2) | 68.3 (7.4) | 66.7 (8.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 9 | 12
  Male | 6 | 12 | 18
Region of Enrollment [Number; unit: participants]
  Australia | 9 | 21 | 30
Ethnicity: Caucasian, Non-Caucasian [Count of Participants; unit: Participants]
  Caucasian | 7 | 17 | 24
  Non-Caucasian | 2 | 4 | 6
Diabetes duration [Median (Inter-Quartile Range); unit: years] | 15.0 [4.0 to 16.0] | 14.0 [11.0 to 18.0] | 14.5 [10.0 to 16.8]
Diabetes Treatment: Mono or dual therapy, Triple or quadruple therapy [Count of Participants; unit: Participants] — Mono or dual therapy refers to treatment with one or two oral hypoglycemic agents.
  Triple or quadruple therapy refers to treatment with three or four oral hypoglycemic agents.
  Participants
    Mono or dual therapy | 5 | 9 | 14
    Triple or quadruple therapy | 4 | 12 | 16
HbA1c [Mean (Standard Deviation); unit: %] | 6.6 (0.8) | 7.0 (0.9) | 6.9 (0.9)
Body Mass Index [Mean (Standard Deviation); unit: kg/m2] | 31.8 (6.3) | 31.2 (5.0) | 31.3 (5.4)
Waist circumference [Mean (Standard Deviation); unit: cm] — Population: Males and Females analysed separately
  cm
    Male: number analyzed (Participants) | 6 | 12 | 18
    Male | 113 (13) | 107 (11) | 109 (13)
    Female: number analyzed (Participants) | 3 | 9 | 12
    Female | 108 (10) | 108 (11) | 108 (10)
Systolic Blood Pressure [Mean (Standard Deviation); unit: mmHg] | 122 (10) | 131 (10) | 128 (11)
Smoking Status: Current, Former, Lifelong non-smoker [Count of Participants; unit: Participants] — Smoking Status: Current refers to those participants currently smoking tobacco products.
  Smoking Status: Former refers to those participants who are not currently smoking but have smoked tobacco products in the past.
  Smoking Status: Lifelong non-smoker refers to those participants who have never smoked tobacco products.
  Participants
    Current | 2 | 0 | 2
    Former | 4 | 6 | 10
    Lifelong non-smoker | 3 | 15 | 18
Alcohol consumption status: Consumer, Abstainer [Count of Participants; unit: Participants] — Participants who reported consuming alcohol are classified as consumers. Participants who reported no alcohol consumption are classified as abstainers.
  Participants
    Consumer | 5 | 17 | 22
    Abstainer | 4 | 4 | 8
Microvascular Complication Status: Present, Absent [Count of Participants; unit: Participants] — Those participants with microvascular complications appear in the "Present" subgroup.
  Those participants without microvascular complications appear in the "Absent" subgroup.
  Participants
    Present | 1 | 8 | 9
    Absent | 8 | 13 | 21

OUTCOME MEASURES:

1. Primary Outcome: Change in the Corrected QT-interval During Nocturnal Hypoglycemia
Description: The nocturnal time period for the study spanned from 11 pm in the evening until 7 am the following morning on two consecutive days. The change in the corrected QT interval during nocturnal hypoglycemia was determined by calculating the difference between the average QTc interval length during periods of hypoglycemia (blood glucose level <3.5 mmol/L) and the average QTc interval length during periods of normoglycemia (blood glucose level >3.5 mmol/L) for the nocturnal time period. The average QTc interval was calculated using an individually optimised correction formula. If the result of average QTc (hypoglycemia) - average QTc (normoglycemia) was positive, the participant experienced QTc prolongation during hypoglycemia. If the result of average QTc (hypoglycemia) - average QTc (normoglycemia) was negative, the participant experienced QTc shortening during hypoglycemia.
Time Frame: Nocturnal time period (2300-0700) during the 48 hours of Holter monitoring
Measure: Count of Participants; unit: Participants
Groups:
- Hypoglycemia Group: While there were nine study participants who experienced hypoglycemia during the entire study period, only eight of those participants experienced hypoglycemia during the nocturnal time period (2300-0700). Six study participants experienced isolated nocturnal hypoglycemia; two study participants experienced both nocturnal and day time hypoglycemia. Hypoglycemia during monitoring was defined as a blood glucose level <3.5mmol/L that was sustained for a minimum of 20 consecutive minutes.
Arm/Group | Hypoglycemia Group
Number analyzed (Participants) | 8
Participants
  QTc prolongation during hypoglycemia | 3
  QTc shortening during hypoglycemia | 5

2. Primary Outcome: Change in Corrected QT Interval During Day Time Hypoglycaemia
Description: The day time period for the study spanned from 7 am in the morning until 11 pm in the evening on two consecutive days. The change in the corrected QT interval during day time hypoglycemia was determined by calculating the difference between the average QTc interval length during periods of hypoglycemia (blood glucose level <3.5 mmol/L) and the average QTc interval length during periods of normoglycemia (blood glucose level >3.5 mmol/L) for the day time period. The average QTc interval was calculated using an individually optimised correction formula. If the result of average QTc (hypoglycemia) - average QTc (normoglycemia) was positive, the participant experienced QTc prolongation during hypoglycemia. If the result of average QTc (hypoglycemia) - average QTc (normoglycemia) was negative, the participant experienced QTc shortening during hypoglycemia.
Time Frame: Day time period (0700-2300) during the 48 hours of Holter monitoring
Measure: Count of Participants; unit: Participants
Groups:
- Hypoglycemia Group: While there were nine study participants who experienced hypoglycemia during the entire study period, only three of those participants experienced hypoglycemia during the day time period (0700-2300). One study participant experienced isolated day time hypoglycemia; two study participants experienced both nocturnal and day time hypoglycemia. Hypoglycemia during monitoring was defined as a blood glucose level <3.5mmol/L that was sustained for a minimum of 20 consecutive minutes.
Arm/Group | Hypoglycemia Group
Number analyzed (Participants) | 3
Participants
  Experienced QTc prolongation during hypoglycemia | 2
  Experienced QTc shortening during hypoglycemia | 1

3. Secondary Outcome: Pearson's Correlation Coefficient of Delta QTc and a Measure of Glucose Variability, MAGE (Mean Amplitude of Glycemic Excursion).
Description: MAGE, a commonly used index of glucose variability, was calculated using data obtained during continuous glucose monitoring. Analysis of correlation between MAGE and delta QTc was undertaken. Please note delta QTc represents the difference between average QTc length during hypoglycemia and average QTc length during normoglycemia.
Time Frame: Nocturnal time period (2300-0700) during the 48 hours of Holter monitoring
Population: The eight study participants who experienced nocturnal hypoglycemia are included in the analysis population.
Measure: Number; unit: Correlation coefficient
Groups:
- Hypoglycemia Group: Those eight participants who experienced hypoglycemia (a Blood Glucose Level <3.5 mmol/L) for a minimum of 20 consecutive minutes during the nocturnal time period (2300-0700) are included in the Hypoglycemia Group for this analysis.
Arm/Group | Hypoglycemia Group
Number analyzed (Participants) | 8
Correlation coefficient | 0.09

4. Secondary Outcome: Mean Amplitude of Glycemic Excursion (MAGE)
Description: The MAGE results (in mmol/L) for the eight participants who experienced nocturnal hypoglycemia are included in the table below.
Time Frame: 48 hours of continuous glucose monitoring
Population: Only those participants who experienced nocturnal hypoglycemia (BGL <3.5 mmol/L for >20 minutes) are included in the analysis population
Measure: Number; unit: mmol/L
Groups:
- Hypoglycemia Group: Those eight participants who experienced hypoglycemia (a Blood Glucose Level <3.5 mmol/L) for a minimum of 20 consecutive minutes during the nocturnal time period (2300-0700) are included in the Hypoglycemia Group for this analysis. The MAGE results for each of the eight participants who experienced hypoglycemia are documented below.
Arm/Group | Hypoglycemia Group
Number analyzed (Participants) | 8
mmol/L
  Participant 1 | 3.9
  Participant 4 | 4.7
  Participant 5 | 3.0
  Participant 10 | 3.9
  Participant 15 | 1.8
  Participant 16 | 3.6
  Participant 19 | 5.7
  Participant 24 | 4.3

5. Secondary Outcome: deltaQTc
Description: deltaQTc is the difference in QTc observed during periods of hypoglycemia and periods of normoglycemia (for those participants who experienced nocturnal hypoglycemia)
Time Frame: Nocturnal time period (2300-0700) during the 48 hours of Holter monitoring
Measure: Number; unit: milliseconds
Groups:
- Hypoglycemia Group: Those eight participants who experienced hypoglycemia (a Blood Glucose Level <3.5 mmol/L) for a minimum of 20 consecutive minutes during the nocturnal time period (2300-0700) are included in the Hypoglycemia Group for this analysis. The results for deltaQTc for each of the eight participants who experienced hypoglycemia are documented below.
Arm/Group | Hypoglycemia Group
Number analyzed (Participants) | 8
milliseconds
  Participant 1 | 10
  Participant 4 | 4
  Participant 5 | -2
  Participant 10 | -6
  Participant 15 | -4
  Participant 16 | -1
  Participant 19 | -8
  Participant 24 | 15

ADVERSE EVENTS:
Arm/Group | Hypoglycemic Group | Normoglycemic Group
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/21
Other Adverse Events (participants affected / at risk) | 9/9 | 0/21
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Hypoglycemic Group (N=9) | Normoglycemic Group (N=21)
Hypoglycemia (Endocrine disorders) | 9 (15) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No